CLINICAL TRIAL: NCT07300371
Title: Intra-oral Evaluation of Force Decay of Pigmented and Transparent Elastomeric Power Chains: A Randomized Clinical Trail.
Brief Title: Intra-oral Evaluation of Force Decay of Pigmented and Transparent Elastomeric Power Chains:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana'a University (Other)
Responsible Party: Principal Investigator, Maha Saleh Mahdi Al-Muntaser, Principal Investigator, Sana'a University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 179
Record Dates: First submitted 2025-11-26; First posted 2025-12-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Orthodontic Treatment; Malocclusion
Keywords: Orthodontic elastomeric power chains or Force decay or Pigmented elastomeric power chains or Transparent elastomeric power chains
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Participant, Investigator
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- Matt gray elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- Matt blue elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- Matt transparent elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- Matt black elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- American orthodocntic gray elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- American orthodontic blue elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- American orthodocntic black elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- American orthodocntic pink elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- American orthodocntic transparent elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- SIA black elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- SIA pink Elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- SIA blue Elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- SIA gray Elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- SIA transparent Elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains
- Matt pink elastomeric power chains (Experimental): EPCs were stretched between the canine bracket hook and the first molar band hook throughout the study period. The delivered force of EPCs was measured using a Dentarum force gauge over 6-week intervals (baseline, after the 1st 24 hours, 1st week, 2nd week, 3rd week, 4th week, 5th week, and 6th week
  Interventions: Other: Matt gray elastomeric power chains; Other: Matt blue elastomeric power chains; Other: Matt pink elastomeric power chains; Other: Matt transparent elastomeric power chains; Other: Matt black elastomeric power chains; Other: American orthodontic gray elastomeric power chains; Other: Americam orthodontic blue elastomeric power chains; Other: Americam orthodontic black elastomeric power chains; Other: Americam orthodontic pink elastomeric power chains; Other: Americam orthodontic transparent elastomeric power chains; Other: SIA pink elastomeric power chains; Other: SIA blue elastomeric power chains; Other: SIA black elastomeric power chains; Other: SIA transparent elastomeric power chains; Other: SIA gray elastomeric power chains

INTERVENTIONS:
Other: Matt gray elastomeric power chains — Matt gray elastomeric power chains is Orthodontic auxiliary/ elastomeric power chains.
Other: Matt blue elastomeric power chains — Orthodontic Auxiliary force generated system
Other: Matt pink elastomeric power chains — Orthodontic Auxiliary force generated system
Other: Matt transparent elastomeric power chains — Orthodontic Auxiliary force generated system
Other: Matt black elastomeric power chains — Orthodontic Auxiliary force generated system
Other: American orthodontic gray elastomeric power chains — Orthodontic Auxiliary force generated system
Other: Americam orthodontic blue elastomeric power chains — Orthodontic Auxiliary force generated system
Other: Americam orthodontic black elastomeric power chains — Orthodontic Auxiliary force generated system
Other: Americam orthodontic pink elastomeric power chains — Orthodontic Auxiliary force generated system
Other: Americam orthodontic transparent elastomeric power chains — Orthodontic Auxiliary force generated system
Other: SIA pink elastomeric power chains — Orthodontic Auxiliary force generated system
Other: SIA blue elastomeric power chains — Orthodontic Auxiliary force generated system
Other: SIA black elastomeric power chains — Orthodontic Auxiliary force generated system
Other: SIA transparent elastomeric power chains — Orthodontic Auxiliary force generated system
Other: SIA gray elastomeric power chains — Orthodontic Auxiliary force generated system

SUMMARY:
This study aimed to evaluate the amount of force decay in pigmented and transparent elastomeric power chains. The principal investigator measured the amount of force decay at 7 intervals using a calibrated Dentaurum force gauge. This study also assessed the associated variables that accelerate the force loss, such as brushing frequency, beverage consumption,mastication, Khat chewing, oral , and tooth movement, . The study outcomes provide evidence-based guidance for selecting elastomeric power chains in routine orthodontic practice.

DETAILED DESCRIPTION:
The study was a split-mouth randomized clinical trial. Four colors (pink, blue, black, and grey) and transparent elastomeric power chains from 3 different companies (American Orthodontic, SIA, and Matt) were evaluated. A total of 96 participants were recruited, and 192 elastomeric power chains were stretched between the canine bracket hook and the molar band hook throughout the study period. The delivered force of elastomeric power chains was assessed and compared among each other using a calibrated Dentarum force gauge over 6-week intervals (baseline, 24 hours, first week, second week, third week, fourth week, fifth week, and sixth week). To further investigate factors influencing force decay (FD), data on tooth movement, mastication side, beverage consumption, brushing frequency, oral hygiene status, and khat chewing were collected using a structured questionnaire to assess their potential impact.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 12-30 years.
2. Patients who are undergoing fixed orthodontic treatment.
3. Orthodontic patients who underwent bilateral extraction protocol in maxillary arch.
4. Patients were in working arch wire 19×25 stainless steel.
5. Patients with moderate anchorage to ensure comparable baseline mechanics.

Exclusion Criteria:

1. Patients indicated for orthognathic treatment.
2. Patients who reported any systemic diseases.
3. Patients with clefts or syndromes.

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2023-11-19 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the force decay of pigmented and transparent elastomeric power chains in a group of orthodontic patients | Baseline and weekly for 6 weeks.
  Measurement of the amount of force decay (in grams) for each elastomeric power chain sample at baseline and at 7 time intervals over 6 weeks using a digital force gauge.

SECONDARY OUTCOMES:
Correlation between force decay and associated variables (tooth movement, masticating side, beverage consumption, brushing frequency, oral hygiene, and khat chewing) | At 6 weeks
  Correlation analysis between force decay values (in grams) and the associated variables collected through a structured questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abdullah Al-Labani, Ph degree, Study Director — Sana'a University,Sana'a,Yemen.
Locations (1):
- Sana'a university, Sanaa, Yemen

IPD SHARING:
Plan to Share IPD: Undecided